CLINICAL TRIAL: NCT04981678
Title: A Prospective, Randomized Trial of the Effect of Buprenorphine Continuation Versus Dose Reduction on Pain Control and Post-Operative Opioid Use
Brief Title: The Effect of Buprenorphine Continuation for Patients With Opioid Use Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was halted prior to accumulating the full number of participants due to difficulty in recruiting study subjects.
Sponsor: MaineHealth (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1688818-1; U54GM115516-06 (NIH)
Record Dates: First submitted 2021-07-08; First posted 2021-07-29 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Buprenorphine Dose Reduction (Other): Patients instructed to reduce buprenorphine to 8mg prior to surgery
  Interventions: Drug: Buprenorphine
- Buprenorphine Full Dose Continuation (Other): Patients instructed to continue taking the full prescribed dose of buprenorphine.
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Patients randomized to this group will reduce their buprenorphine dose prior to surgery.
  Arms: Buprenorphine Dose Reduction
Drug: Buprenorphine — Patients randomized to this group will continue their buprenorphine at the full prescribed dose.
  Arms: Buprenorphine Full Dose Continuation

SUMMARY:
There is limited guidance on the optimal management of buprenorphine perioperatively and both buprenorphine discontinuation and continuation are acceptable standards of care. Buprenorphine continuation at low analgesic dosing is also accepted, however is not provided as a potential treatment strategy by the Substance Abuse and Mental Health Services Administration (SAMHSA). There is the risk of inadequate pain control necessitating opioid escalation when buprenorphine is continued. Preliminary clinical observations support buprenorphine continuation at low analgesic doses (8mg) as it adequately facilitates postoperative pain management without interrupting opioid use disorder (OUD) treatment, however to date, no prospective trial has investigated this treatment strategy in comparison to full dose buprenorphine continuation. Since optimal perioperative dosing strategies remain unknown, the purpose of this study is to investigate if buprenorphine continuation at analgesic dosing is superior to full dose buprenorphine continuation in individuals presenting for elective surgery.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether buprenorphine continuation at analgesic dosing is superior to full dose buprenorphine continuation in individuals presenting for elective surgery. Adults scheduled for elective surgery who are taking ≥12mg buprenorphine for OUD treatment will be eligible for this study. Enrolled participants will be randomized to receive either a reduced analgesic dose of buprenorphine (8mg) or to continue buprenorphine on the day of surgery without dose reduction. The primary outcome of interest is postoperative pain scores. The secondary outcomes of interest are opioid consumption, opioid dispensing up to 30 days following the surgical procedure and OUD related symptoms, including opioid withdrawal, cravings and relapse. The investigators hypothesis is that there will be a clinically significant increase in pain scores when buprenorphine is continued in full compared to when it is continued at a lower analgesic dose. Clinical significance will be defined as a difference in composite pain scores of greater than 20% between groups. The investigators also hypothesize that opioid consumption and opioid dispensing will be greater with full dose buprenorphine continuation compared to low-dose continuation.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and older
* American Society of Anesthesia health class I-III
* Currently taking buprenorphine formulation equivalent to 12mg or greater for at least 30 days for treatment of Opioid Use Disorder
* Scheduled for surgery at Maine Medical Center for a procedure with a greater than 4/10 pain intensity is expected on post-op day one.

Exclusion Criteria:

* unable to consent to the study
* currently pregnant
* current major medical illness that could limit the ability to utilize medications within our protocol driven multimodal analgesic plan (e.g. cancer, severe end-stage organ disease, or dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aurora Quaye, MD, Principal Investigator — Maine Medical Center; Spectrum Healthcare Partners
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (5.3) | 40.5 (5.7) | 40.6 (50.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Current buprenorphine dose [Median (Full Range); unit: mg] | 15 [12 to 20] | 16 [16 to 24] | 16 [12 to 24]

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Scores: 24 Hours After Surgery
Description: Highest, average, and lowest pain scores will be evaluated using the Numerical Rating Scale of 0 (no pain) -10 (worst pain)
Time Frame: 24 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale (NRS pain scale)
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Number analyzed (Participants) | 6 | 6
score on a scale (NRS pain scale)
  Average | 7.2 (1.5) | 5.8 (2.4)
  Lowest | 6.0 (2.4) | 4.5 (2.7)
  Highest | 8.3 (1.4) | 7.4 (2.8)

2. Primary Outcome: Post-operative Pain Scores: 48 Hours After Surgery
Description: as for outcome 1
Time Frame: 48 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale (NRS)
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Number analyzed (Participants) | 6 | 6
score on a scale (NRS)
  Average | 6.8 (2.5) | 5.4 (1.6)
  Lowest | 6.2 (2.5) | 2.8 (0.8)
  Highest | 7.8 (2.3) | 7.7 (2.1)

3. Primary Outcome: Post-operative Pain Scores: 72 Hours After Surgery
Description: as for outcome 1
Time Frame: 72 hours after surgery
Measure: Mean (Standard Deviation); unit: score on a scale (NRS)
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Number analyzed (Participants) | 6 | 6
score on a scale (NRS)
  Average | 6.6 (1.6) | 5.1 (2.3)
  Lowest | 5.2 (1.6) | 4.1 (2.5)
  Highest | 7.4 (1.9) | 6.1 (2.4)

4. Secondary Outcome: Opioid Consumption
Description: All opioids consumed through 72 hours after surgery combined into mean morphine equivalents
Time Frame: 3 days post-op
Measure: Mean (Full Range); unit: morphine milligram equivalents (MME)
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Number analyzed (Participants) | 6 | 6
morphine milligram equivalents (MME) | 37.25 [0 to 140] | 41.43 [0 to 320]

5. Secondary Outcome: Opioid Dispensing
Description: Prescriptions filled for the patient in the Prescription Awareness Tool
Time Frame: 30 days following surgery
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Number analyzed (Participants) | 6 | 5
morphine milligram equivalents | 262 [0 to 915] | 308 [0 to 519]

6. Secondary Outcome: Opioid Withdrawal
Description: Withdrawal symptoms as measured by the Clinical Opioid Withdrawal Scale (COWS, scores can range from 0-48 [5-12 mild; 13-24, moderate; 25-36, moderately severe; >36, severe withdrawal)
Time Frame: 1-3 hours prior to surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Number analyzed (Participants) | 6 | 6
Participants
  less than 5 on the COWS scale | 5 | 5
  5-12 on the COWS scale, mild withdrawal | 1 | 1

7. Secondary Outcome: Opioid Cravings
Description: Measured by the Opioid Craving Scale (OCS); scale ranges from 0-30 with higher scores indicating higher levels of cravings
Time Frame: 1-3 hours prior to surgery
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Number analyzed (Participants) | 6 | 6
score on a scale | 2.17 [0 to 9] | 2 [0 to 6]

8. Secondary Outcome: Opioid Cravings
Description: as for outcome 7
Time Frame: 30 days following surgery
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Number analyzed (Participants) | 6 | 5
score on a scale | 0.67 [0 to 4] | 3 [0 to 13]

9. Secondary Outcome: Opioid Misuse
Description: Measured by the Current Opioid Misuse Measure ((COMM); scores can range from 0-68, scores of 9 or lower indicates a low risk of opioid misuse or abuse, scores higher than 9 indicate a high risk)
Time Frame: 1-3 hours prior to surgery
Measure: Mean (Full Range); unit: score on a scale (COMM)
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Number analyzed (Participants) | 6 | 6
score on a scale (COMM) | 2.83 [0 to 10] | 7 [0 to 15]

10. Secondary Outcome: Opioid Misuse
Description: as for outcome 9
Time Frame: 30 days following surgery
Measure: Mean (Full Range); unit: score on a scale (COMM)
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Number analyzed (Participants) | 6 | 5
score on a scale (COMM) | 3.33 [0 to 10] | 8 [1 to 18]

11. Secondary Outcome: Opioid Relapse
Description: Patient reported use of non-prescribed opioids
Time Frame: 30 days following surgery
Measure: Number; unit: number of patients reporting relapse
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
Number analyzed (Participants) | 6 | 5
number of patients reporting relapse | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Buprenorphine Dose Reduction | Buprenorphine Full Dose Continuation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Early termination due to low enrollment; limited data analysis performed because of the small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/78/NCT04981678/Prot_SAP_000.pdf